CLINICAL TRIAL: NCT03929601
Title: Rituximab-pvvr and Abatacept vs Rituximab-pvvr Alone in New Onset Type 1 Diabetes
Acronym: TN25
Status: Active, not recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: National Institute of Diabetes and Digestive and Kidney Diseases (NIDDK) (NIH)
Collaborators: National Institutes of Health (NIH) (NIH)
Responsible Party: Sponsor
Allocation: Randomized | Model: Sequential | Masking: Triple | Purpose: Treatment
Other Study IDs: Rituximab-pvvr and Abatacept; UC4DK117009 (NIH)
Record Dates: First submitted 2018-05-16; First posted 2019-04-29 (Actual); Last update posted 2025-07-02 (Actual); Status verified 2025-06

CONDITIONS: Type 1 Diabetes Mellitus
MeSH Terms: conditions — Diabetes Mellitus, Type 1 | interventions — Abatacept; Injections

STUDY DESIGN:
Intervention Model Description: This protocol will enroll 74 participants who will be treated with a course of rituximab-pvvr (weekly infusion for 4 weeks), followed by treatment with abatacept or placebo starting at 4 months after initial rituximab-pvvr treatment and continuing to month 24. The abatacept/placebo treatment will be self-administered by participants (or their families/guardians, where most appropriate, particularly with pediatric participants) weekly for 20 months. Rituximab-pvvr will be given by IV infusion over at least 3 hours, at a dose of 375mg/m2 on four visits each one week apart, starting at Week 0 of the study. Abatacept/placebo will be given by a subcutaneous formulation weekly for 20 months, beginning at Week 16 (Month 4) of the study. Dosing will be determined by weight: Up to 25 kg: 50 mg (0.4 mL); 25 to <50 kg receive 87.5 mg (0.7 mL), and > 50 kg receive 125 mg (1.0 mL).
Who Masked: Participant, Care Provider, Investigator
Masking Description: This study is double blinded.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: Yes

ARMS (2):
- Rituximab-pvvr followed by Abatacept (Active Comparator): Rituximab-pvvr will be given by IV infusion over at least 3 hours, at a dose of 375mg/m2 on four visits each one week apart, starting at Week 0 of the study.
  Abatacept will be given by a subcutaneous formulation weekly for 20 months, beginning at Week 16 (Month 4) of the study. Dosing will be determined by weight: Up to 25 kg: 50 mg (0.4 mL); 25 to <50 kg receive 87.5 mg (0.7 mL), and > 50 kg receive 125 mg (1.0 mL).
  Interventions: Drug: Rituximab-pvvr; Drug: Abatacept
- Rituximab-pvvr followed by Placebo (Placebo Comparator): Rituximab-pvvr will be given by IV infusion over at least 3 hours, at a dose of 375mg/m2 on four visits each one week apart, starting at Week 0 of the study.
  Placebo will be given by a subcutaneous isotonic saline formulation weekly for 20 months, beginning at Week 16 (Month 4) of the study. Dosing will be match to active comparator, determined by weight: Up to 25 kg: 0.4 mL; 25 to <50 kg rec 0.7 mL, and > 50 kg receive 1.0 mL.
  Interventions: Drug: Rituximab-pvvr; Drug: Sterile Sodium Chloride

INTERVENTIONS:
Drug: Rituximab-pvvr — All participants will receive Rituximab-pvvr dosing from Week 1 to Week 4 of the trial. Rituximab-pvvr will be given by IV infusion over at least 3 hours, at a dose of 375mg/m2 on four visits each one week apart.
  Other Names: Ruxience
Drug: Abatacept — Participants in the active drug arm will receive initial Abatacept dosing at Week 16 of trial. Abatacept will be given by a subcutaneous (SC) formulation weekly for 20 months, and dosing be will determined according to weight: Up to 25 kg: 50 mg (0.4 mL); 25 to <50 kg receive 87.5 mg (0.7 mL), and > 50 kg receive 125 mg (1.0 mL).
  Other Names: Orencia
  Arms: Rituximab-pvvr followed by Abatacept
Drug: Sterile Sodium Chloride — Participants in the placebo arm will receive initial placebo injection at Week 16 of trial. Saline Placebo will be given by a subcutaneous (SC) formulation weekly for 20 months, and dosing volume be will determined according to weight to match active comparator: Up to 25 kg: 0.4 mL; 25 to <50 kg receive 0.7 mL and > 50 kg receive 1.0 mL.
  Other Names: 0.9% Sodium Chloride Water for Injection
  Arms: Rituximab-pvvr followed by Placebo

SUMMARY:
The study is a two-arm, multicenter, double-blinded clinical trial testing sequential therapy with rituximab-pvvr followed by abatacept versus rituximab-pvvr alone in new onset T1D. The primary objective is to test whether the C-peptide response to a 2-hour mixed meal tolerance test, will be improved in participants with new onset T1D who are treated with Abatacept after Rituximab-pvvr compared to those treated with Rituximab-pvvr and placebo 24 months after enrollment.

DETAILED DESCRIPTION:
This is a two-arm, double-blind, multicenter clinical trial testing sequential therapy with rituximab-pvvr followed by abatacept versus rituximab-pvvr alone in individuals with new onset T1D to determine whether rituximab-pvvr followed by abatacept results in an improvement in the AUC C-Peptide during a MMTT compared to Rituximab-pvvr alone at 24 months. Additional aims will compare the safety, tolerability in the two treatment arms as well as other clinical metabolic measures: exogenous insulin use, hemoglobin A1c, time in range from continuous glucose monitors, and severe hypoglycemia. Exploratory studies will assess changes in immune markers.

ELIGIBILITY:
Inclusion Criteria:

1. Age ≥ 8 and ≤ 45 years old at time of signing informed consent.
2. Fulfill the ADA criteria for diagnosis of T1D within 100 days of randomization.
3. Must be willing to provide informed consent or assent with a parent or legal guardian providing informed consent if < 18 years of age.
4. Positive for at least one islet cell autoantibody; GAD65A, mIAA (if obtained within 10 days of the onset of insulin therapy), IA-2A, ICA, or ZnT8A
5. Must have stimulated C-peptide of ≥0.2 pmol/mL measured during mixed-meal tolerance test (MMTT) conducted at least 21 days after the diagnosis of diabetes.
6. Enrollees must be willing to comply with intensive diabetes management.
7. Body weight must be ≥ 20.0 kg for study agent administration.
8. Subjects who are CMV and/or EBV seronegative at screening must be CMV and/or EBV PCR negative and may not have had signs or symptoms of a CMV and/or EBV compatible illness prior to randomization.
9. Female participants with reproductive potential must have a negative pregnancy test at screening and be willing to avoid pregnancy for the duration of treatment and until 3 months after the last dose of Abatacept. Female participants with reproductive potential who are sexually active will be instructed to use a highly effective contraceptive method until one year after the last dose of rituximab-pvvr.
10. Male participants of reproductive age must use an adequate contraceptive method for the duration of rituximab-pvvr treatment and 12 months following the last dose of rituximab-pvvr.
11. The following additional inclusion criteria regarding vaccines must be met:

    1. More than 4 weeks from immunization with a live viral vaccine
    2. Be up to date on all recommended vaccinations based on age of subject*
    3. Receive non-live influenza vaccination at least 2 weeks prior to randomization when vaccine for the current or upcoming flu season is available
    4. Willingness to forgo vaccines (other than killed influenza) during the 6 months after the rituximab-pvvr treatment period
12. Participants must be willing to practice public health prevention measures such as social distancing, masking, and good hand hygiene, and/or receive therapeutics such as monoclonal antibodies and antivirals as directed by the study and recommended by local health authorities to prevent SARS-Cov-2 infection.
13. Willing to wear a continuous glucose monitoring device for a minimum of 10 days every 6 months

    * Adult participants must be fully immunized. Pediatric subjects who have not completed their primary vaccination schedule must receive all vaccinations allowable per local public health immunization guidelines for their current age prior to study drug delivery. HPV vaccine may be initiated and/or series completion delayed until after completion of study drug in both adult and pediatric participants. Any remaining vaccinations should be given and continue per the schedule at least 6 months after rituximab-pvvr is administered. For COVID-19 vaccination, all participants will be strongly encouraged to be up-to-date with COVID-19 vaccine(s) as indicated by country-specific guidelines at least 2 weeks prior to randomization.

Exclusion Criteria:

1. One or more screening laboratory values as stated:

   1. Leukocytes <3,000/μL
   2. Neutrophils <1,500/μL
   3. Lymphocytes <800/μL
   4. Platelets <100,000/μL
   5. Hemoglobin <6.2 mmol/L (10.0 g/dL)
   6. Potassium >5.5 mmol/L or <3.0 mmol/L
   7. Sodium >150 mmol/L or <130 mmol/L
   8. AST or ALT ≥ 2.5 times the upper limits of normal
   9. Total bilirubin ≥ 1.5 times upper limit of normal, except in the case of Gilbert's disease
2. History of immune deficiency
3. Current or ongoing use of non-insulin pharmaceuticals that affect glycemic control within 7 days of screening visit.
4. Chronic active infection other than localized skin infections.
5. Have active signs or symptoms of acute infection at the time of randomization.
6. Have IgG and/or IgM levels below the normal reference ranges.
7. Positive PPD, interferon gamma release assay (IGRA) or history of previous treatment for TB.
8. Vaccination with a live virus within 4 weeks prior to initiating study treatment.
9. A history of confirmed infectious mononucleosis within the 3 months prior to initiating study treatment, as documented by EBV serology (EBV VCA-IgM and VCA-IgG; PCR would be confirmatory).
10. Laboratory evidence of current or past HIV or Hepatitis B or active Hepatitis C infection.
11. Be currently pregnant, lactating or anticipate pregnancy within 14 weeks of the last study drug administration (Visit 15).
12. Chronic use of oral or inhaled steroids or other immunosuppressive agents.
13. Known and untreated hypothyroidism or active Graves' disease at randomization.
14. History of malignancy.
15. Prior treatment with active study agent from a previous T1D clinical trial.*
16. Have had previous clinical use of Tzield (Teplizumab) not part of a T1D treatment study.
17. Any laboratory abnormality or condition that, in the opinion of the investigator, would interfere with the study conduct or the safety of the participant.

    * Study drug exposure may be reviewed by the TrialNet Eligibility and Events Committee and determination will be made as to whether subjects can be considered eligible for this study based on agent, length of time since exposure, duration of treatment, durability of effect, and potential for lingering immunomodulation.

Ages: 8 Years to 45 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 74 (Actual)
Dates: Start 2023-10-30 (Actual); Primary Completion 2027-03-31 (Estimated); Study Completion 2029-03-31 (Estimated)

PRIMARY OUTCOMES:
C-Peptide Response to 2-hr MMTT at 24 months post-randomization | 48-months from Day 0
  The primary objective is to test whether the C-peptide response to a 2-hour mixed meal tolerance test, will be improved in participants with new onset T1D who are treated with Abatacept after Rituximab compared to those participants treated with Rituximab and placebo 24 months after enrollment.

SECONDARY OUTCOMES:
C-peptide AUC Means | Day 0 and every 6 months to trial end (up to 4 years)
  C-peptide AUC Mean at 0, 6, 12, 18, 24, 30, 36, 42 and 48 months using the ANCOVA model.
Analysis of changes in immune responses to known diabetes antigens and a neoantigen over time by treatment group | Day 0, month 2, 4, 5, 6, 12, 13, 18, 24, 25, 30, and 36
  Analysis of changes in immune responses to known diabetes antigens and a neoantigen. The investigators will compare the effects of drug treatments on the titers of autoantibodies: anti-insulin, anti-GAD65, anti-IA-2, anti-ZnT8. The investigators will also compare the effects of drug treatments on the response to Keyhole Limpet Hemocyanin (KLH) for which standardized immunological responses have been characterized.

CONTACTS AND LOCATIONS:
Overall Officials: Stephen Gitelman, MD, Study Chair — Type 1 Diabetes TrialNet; Kevan Herold, MD, Study Director — Type 1 Diabetes TrialNet Chairman; Daniel Moore, MD, Study Chair — Type 1 Diabetes TrialNet
Locations (19):
- United States (17):
  - Childrens Hospital of Orange County, Orange, California
  - Stanford University, Palo Alto, California
  - University of California San Francisco, San Francisco, California
  - Barbara Davis Center for Childhood Diabetes, Aurora, Colorado
  - Yale University, New Haven, Connecticut
  - University of Florida, Gainesville, Florida
  - University of Miami, Maimi, Florida
  - Indiana University - Riley Hospital for Children, Indianapolis, Indiana
  - The Children's Mercy Hospital, Kansas City, Kansas
  - Joslin Diabetes Center, Boston, Massachusetts
  - University of Minnesota, Minneapolis, Minnesota
  - Columbia University, New York, New York
  - University of Pittsburg, Pittsburgh, Pennsylvania
  - Sanford Children's Specialty Clinic, Sioux Falls, South Dakota
  - Vanderbilt Eskind Diabetes Center, Nashville, Tennessee
  - University of Texas Southwestern, Dallas, Texas
  - Benaroya Research Institute, Seattle, Washington
- Australia (2):
  - Queensland Children's Hospital, South Brisbane, Queensland
  - Walter and Eliza Hall Institute of Medical Research, Melbourne, Victoria

IPD SHARING:
Plan to Share IPD: Yes

REFERENCES:
- [Derived] Ajmal N, Bogart MC, Khan P, Max-Harry IM, Healy AM, Nunemaker CS. Identifying Promising Immunomodulators for Type 1 Diabetes (T1D) and Islet Transplantation. J Diabetes Res. 2024 Dec 20;2024:5151171. doi: 10.1155/jdr/5151171. eCollection 2024. PMID 39735417
- See also: Study Sponsor Website — http://www.trialnet.org/